CLINICAL TRIAL: NCT07204028
Title: Corpus Luteum Doppler in Prediction of First Trimester Pregnancy Outcome
Brief Title: Early Pregnancy Ultrasound Parameters Including Corpus Luteum Doppler in Prediction of First Trimester Pregnancy Outcome in Spontaneous Pregnancies.
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mostafa Mohammed Refaay El shemy, Assistant professor at obstetrics and gynecology department, Cairo University
Other Study IDs: Corpus luteum Doppler
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Fetal Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The synthesis of progesterone by corpus luteum is extremely important for the maintenance of normal pregnancy in the first seven weeks. Similarly, the production of progesterone by the placental syncytiotrophoblast increases progressively during the first weeks of gestation, so that in eight and a half weeks the placenta and corpus luteum contribute in equal amounts of progesterone. However, from the eighth week, the placental contribution is sufficient to maintain gestation. Angiogenesis in the corpus luteum occurs under physiologic circumstances in each menstrual cycle and functionally is very important for maintenance of early pregnancy. This role implies a potential correlation between abnormal function of corpus luteum and possible abnormal pregnancy including abortion. Using color Doppler sonography, it was feasible to distinguish the ovary containing an active corpus luteum from the inactive ovary. The technique is simple to use, and the results are displayed obviously (Abd-elfatah & Megahed, 2020). 6 and

DETAILED DESCRIPTION:
Gestational sac (GS), yolk sac (YS), crown-rump length (CRL), and heart rate (HR) and corpus luteum Doppler are the parameters measured to evaluate early pregnancy. Deviations in the ultrasound parameters have been alternatively investigated to predict first trimester pregnancy loss. The amniotic sac, which becomes visible at the beginning of the 7th week of gestation, is normally not contemplated in the prediction models, however it assists in dating a pregnancy correctly (Detti et al., 2020).

The aim of this study is to evaluate gestational sac diameter (GSD), yolk sac diameter (YSD), heart rate (HR), CRL and corpus luteum Doppler at 6-12 gestational weeks (GW) as predictors of first trimester outcome.

ELIGIBILITY:
Inclusion Criteria:

* The age of women in the studied population was up to 40 years.
* Live singleton pregnancy with gestational age 6-9 gestational weeks.
* Patients with threatened miscarriage were included.

Exclusion Criteria:

* Ectopic pregnancy.
* Multiple pregnancies.
* Vesicular mole.
* Miscarriage in first visit.
* Fetal anomaly.
* Known uterine anomalies.
* Significant pre-pregnancy maternal diseases (e.g., hypertension - diabetes mellitus-systemic lupus) or known thrombophilia (e.g., antiphospholipid syndrome).

Max Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant female aged less than 40 years at 6-12 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
New predictors of first trimester pregnancy outcome | 6 months
  Evaluation of corpus luteum Doppler as predictor of first trimester outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo University, Giza, Cairo Governorate, Egypt